CLINICAL TRIAL: NCT04420273
Title: Targeted Melanoma Detection With Skin Self-examination: Leveraging the Mammogram Encounter
Brief Title: Targeted Melanoma Detection With Skin Self-Examination During COVID-19 Restricted Physician Access
Acronym: TMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, Research Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU00212165
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: Randomized Control Clinical Trial Arm 1: SSE educational intervention with optional physician supervised non-invasive adhesive patch-based home sample collection of a concerning mole for genomic analysis Arm 2: Active control
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSE educational intervention (Experimental): Women participants receive a SSE brochure and three monthly reminders to perform SSE. In the second month, women select goals for SSE.
  Interventions: Behavioral: SSE educational intervention
- Active control: Healthy Living (Active Comparator): Women participants receive a Healthy Living brochure and three monthly reminders to perform the following activities of healthy living: get quality sleep, walk briskly for 30 min, eat 5 servings of fruits and vegetables a day. In the second month, women select goals for healthy living.
  Interventions: Behavioral: Active control:Healthy Living

INTERVENTIONS:
Behavioral: SSE educational intervention — Women participants receive a SSE brochure and three monthly reminders to perform SSE. In the second month, women select goals for SSE.
  Arms: SSE educational intervention
Behavioral: Active control:Healthy Living — Women participants receive a Healthy Living brochure and three monthly reminders to perform the following activities of healthy living: get quality sleep, walk briskly for 30 min, eat 5 servings of fruits and vegetables a day. In the second month, women select goals for healthy living.
  Arms: Active control: Healthy Living

SUMMARY:
The purpose of this study is to reduce melanoma mortality by improving early detection of melanoma with skin self-examination (SSE) among people who self-identify as being at risk and seek care for a concerning mole. Because women are more likely than men to perform SSE, women who are engaged in health promotion by having a recent screening mammogram are the focus of this research. Self-management of melanoma detection with SSE depends on ready access to dermatologists when a concerning mole is detected. In March 2020, the Illinois stay at home order (COVID-19) prohibited non-essential health care, including screening mammography and dermatology office-based care, and both are expected to remain limited until fall 2020. This submission explores a) the effectiveness of targeted melanoma detection (TMD) among women, who identify their risk of having a melanoma, learn to perform SSE, and perform SSE, and b) the effectiveness of adhesive patch-based home sample collection for genomic analysis to rule out melanoma in moles identified by women (who received the intervention) as concerning will be explored.

DETAILED DESCRIPTION:
The proposed work will assess the effectiveness of targeted melanoma detection (TMD) with SSE education delivered remotely to women who had a screening mammogram. The effect of TMD with SSE education will be assessed with a randomized control trial among women served by Northwestern Medicine in rural, suburban and metropolitan communities. Women who identify concerning moles will choose among three options: a) watch the mole to see if the border, color or diameter of the mole changes b) send a picture of the mole to the PI for consideration of mole self-sampling, or c) make an appointment with my healthcare provider to check the mole. As required a physician will supervise women, who will perform non-invasive mole self-sampling with non-invasive adhesive patches for genomic analysis of the concerning pigmented lesion (mole). If the genomic analysis suggests that the concerning mole may be a melanoma, then the recommendation will be to have the mole biopsied.The effectiveness of acquired samples suggestive of melanoma will be examined by the obtaining the pathology reports of biopsied moles. Health care providers' (HCPs) clinical/pathologic assessment of concerning moles will be identified in the Northwestern Medicine electronic health record (EHR) system.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (aged 18 and older) with no upper age limit, who had a screening mammogram from January 1, 2019 to February 28, 2020.
* Able to read English
* Vision enough to read a newspaper
* Self-perception of their potential melanoma risk
* Willing to perform SSE either alone or with a skin check partner
* Willing to complete monthly surveys for 3 months and receive monthly text messages to personal mobile phone
* Have home Internet access and phone with ability to take a picture of a mole
* Have access to Federal Express or US Postal Service Express Mail to send mole self-sampling kits
* Willing to allow the research team access to their electronic health record to abstract physician assessment of concerning moles, biopsy results and treatment
* Willing to provide up-to-date email address, mailing address and telephone number

Inclusion criteria of skin check partner, who may be a man or a woman, to have mole self-sampled

* Male or female over the age of 18 years
* Able to read English
* Vision enough to read a newspaper

Exclusion Criteria:

* Male
* Female under the age of 18
* Unable to read English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation as a woman
Enrollment: 1000 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: June K Robinson, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robinson JK, Reavy R, Mallett KA, Turrisi R. Remote partner assisted skin self-examination skills training of melanoma survivors and their partners. Australas J Dermatol. 2019 Feb;60(1):e80-e82. doi: 10.1111/ajd.12877. Epub 2018 Jul 10. No abstract available. PMID 30773613
- [Background] Robinson JK, Wayne JD, Martini MC, Hultgren BA, Mallett KA, Turrisi R. Early Detection of New Melanomas by Patients With Melanoma and Their Partners Using a Structured Skin Self-examination Skills Training Intervention: A Randomized Clinical Trial. JAMA Dermatol. 2016 Sep 1;152(9):979-85. doi: 10.1001/jamadermatol.2016.1985. PMID 27367303

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SSE Educational Intervention | Active Control: Healthy Living
Started | 501 | 499
Completed | 390 | 414
Not Completed | 111 | 85

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SSE Educational Intervention | Active Control: Healthy Living | Total
Number analyzed (Participants) | 494 | 495 | 989
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 494 | 495 | 989
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47.0 [41.2 to 54.0] | 47.0 [41.0 to 53.3] | 47.0 [41.1 to 53.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 494 | 495 | 989
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 36 | 73
  Not Hispanic or Latino | 457 | 459 | 916
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 485 | 480 | 965
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 3 | 6 | 9
skin type [Count of Participants; unit: Participants]
  I (always sunburn, never tan) | 29 | 22 | 51
  II (usually sunburn, tan minimally) | 213 | 230 | 443
  III (sometimes sunburn, tan moderately) | 216 | 200 | 416
  IV(rarely sunburn, tan deeply) | 36 | 43 | 79

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed SSE at Specified Time Points
Description: Self-reported performance of SSE, a custom scale with the frequency and extent of SSE is completed in an online monthly survey
Time Frame: 90 days
Population: Home sample collection arm participants were randomized into arm 1 at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | SSE Educational Intervention | Active Control: Healthy Living
Number analyzed (Participants) | 494 | 495
Participants
  baseline ever perform SSE | 217 | 242
  1-mo perform SSE | 475 | 238
  2-mo perform SSE | 355 | 228
  3-mo perform SSE | 348 | 211
Statistical Analysis 1: Comparison: SSE Educational Intervention vs Active Control: Healthy Living; 1-month survey; Test type: Other; p < 0.001, McNemar; McNemar's chi-square with continuity correction
Statistical Analysis 2: Comparison: SSE Educational Intervention vs Active Control: Healthy Living; 2- months; Test type: Other; p < 0.001, McNemar; McNemar's chi-square with continuity correction
Statistical Analysis 3: Comparison: SSE Educational Intervention vs Active Control: Healthy Living; 3-months; Test type: Other; p < 0.001, McNemar; McNemar's chi-square with continuity correction

2. Primary Outcome: Number of Participants Who Identified Concerning Moles at Specified Time Points
Description: Self-reported identification of concerning mole identified by user assigning scores to the border,color and diameter of the mole. A validated scoring system is used to categorize the border, color and diameter as 1 if normal, 2 if not sure, and 3 if abnormal.The sum of the scores indicates if the mole is concerning (sum of 3= benign, stop checking the mole; sum of 4- 7 monitor the mole for change in the next month; sum of 8-9 = concerning mole make an appointment to see a physician.
Time Frame: 90 days
Population: While 494 participants were randomized to receive the intervention, only 278 participants found a concerning mole. Similarly 495 participants were randomized to the active control arm, but only 144 identified a concerning mole. Thus the number analyzed in each arm is limited to the number of participants identifying a concerning mole.
Measure: Count of Participants; unit: Participants
Arm/Group | SSE Educational Intervention | Active Control: Healthy Living
Number analyzed (Participants) | 278 | 144
Participants
  Made physician appointment | 39 | 107
  Followed mole for change | 239 | 7
  stopped SSE | 0 | 30
Statistical Analysis 1: Comparison: SSE Educational Intervention vs Active Control: Healthy Living; Test type: Other; p < 0.001, Chi-squared

3. Secondary Outcome: Participants' Reported Skin Self-examination Anxiety
Description: Self-reported responses to 6 items, each with a 5-point Likert scale (range 6-30) higher score= more anxiety, a worse outcome
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SSE Educational Intervention | Active Control: Healthy Living
Number analyzed (Participants) | 390 | 414
units on a scale
  Baseline | 6.4 (0.05) | 6.4 (0.05)
  Follow-up month 3 | 6.6 (0.05) | 6.6 (0.05)
Statistical Analysis 1: Comparison: SSE Educational Intervention vs Active Control: Healthy Living; Test type: Other; p < 0.1, Chi-squared

4. Secondary Outcome: Participants' Confidence Performing Mole Checks
Description: Self-reported responses to 7 items, each with a 5-point Likert scale (range 7-35) higher score = greater confidence (better outcome).
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SSE Educational Intervention | Active Control: Healthy Living
Number analyzed (Participants) | 390 | 414
units on a scale
  Baseline | 9.3 (0.05) | 9.3 (0.05)
  Follow-up-3 month | 11.6 (0.05) | 10.0 (0.05)
Statistical Analysis 1: Comparison: SSE Educational Intervention vs Active Control: Healthy Living; Test type: Other; p < 0.001, Chi-squared

5. Secondary Outcome: Clinical Diagnosis of Participants Having Any Physician Visits for Concerning Moles
Description: Electronic medical record review of physician's clinical diagnosis of concerning mole during the 3 months of the study and for 2 subsequent months
Time Frame: 5 months
Measure: Number; unit: participants
Arm/Group | SSE Educational Intervention | Active Control: Healthy Living
Number analyzed (Participants) | 39 | 107
participants
  Clinical diagnosis benign | 14 | 93
  Clinical diagnosis atypical nevus | 15 | 9
  Clinical diagnosis melanoma | 10 | 5
Statistical Analysis 1: Comparison: SSE Educational Intervention vs Active Control: Healthy Living; Test type: Other; p < 0.001, Chi-squared

6. Secondary Outcome: Pathologic Diagnosis of Concerning Moles
Description: Electronic medical record review of pathologic diagnosis of biopsied moles that participants identified as concerning
Time Frame: 5 months
Population: all participants in arm 3 had benign moles on the home sample collected
Measure: Number; unit: participants
Arm/Group | SSE Educational Intervention | Active Control: Healthy Living
Number analyzed (Participants) | 22 | 14
participants
  benign nevus | 0 | 1
  atypical nevus | 13 | 6
  melanoma stage 0 | 5 | 3
  melanoma stage 1A | 4 | 3
  melanoma stage 1B | 0 | 1
Statistical Analysis 1: Comparison: SSE Educational Intervention vs Active Control: Healthy Living; Test type: Other; p = 0.459, Chi-squared
Statistical Analysis 2: Comparison: SSE Educational Intervention vs Active Control: Healthy Living; Test type: Superiority; p < 0.001, Chi-squared

7. Secondary Outcome: Biopsy Performed
Description: EMR review of physician performing a biopsy on a concerning mole identified by the participant, percentage of biopsies performed
Time Frame: 5 months
Population: percentage of participants having a biopsy of a concerning mole
Measure: Number; unit: percentage of participants having a biop
Arm/Group | SSE Educational Intervention | Active Control: Healthy Living
Number analyzed (Participants) | 39 | 107
percentage of participants having a biop | 56.4 | 13.1
Statistical Analysis 1: Comparison: SSE Educational Intervention vs Active Control: Healthy Living; Test type: Other; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: two months after completing final 3-month survey of study
Arm/Group | SSE Educational Intervention | Active Control: Healthy Living
All-Cause Mortality (participants affected / at risk) | 0/494 | 0/495
Serious Adverse Events (participants affected / at risk) | 0/494 | 0/495
Other Adverse Events (participants affected / at risk) | 0/494 | 0/495

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT04420273/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-31): https://cdn.clinicaltrials.gov/large-docs/73/NCT04420273/ICF_001.pdf